CLINICAL TRIAL: NCT03848338
Title: Evaluation of Intra and Post-operative Electrocochleography for the Monitoring of Residual Hearing
Brief Title: Electrocochleography Function for Monitoring Residual Hearing
Acronym: ECochG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 214480
Record Dates: First submitted 2019-02-08; First posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Hearing Loss, Cochlear
Keywords: Cochlear Implant; Electrocochleography
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Pilot Group (Other): Intra and Post-operative Electrocochleography
  Interventions: Procedure: Electrocochleography

INTERVENTIONS:
Procedure: Electrocochleography — Electrocochleography measurement Intra-operatively and Post-operatively at follow-up appointments along with correlative measurements (Impedance, eCAP, PTA, Speech)

SUMMARY:
This trial is a pilot study to assess the feasibility of using Electrocochleography recorded from a cochlear implant intra-operatively in real time to monitor the progress of its insertion. Correlation between:

1. Observed changes in this signal during surgery and residual hearing loss post-operatively and
2. Recordings of this signal post-operatively and actual pure tone audiometry results will also be assessed.

DETAILED DESCRIPTION:
Cochlear Implants (CIs) can provide deaf individuals the ability to hear. CIs are electronics packages inserted into the cochlea (hearing organ). An external processor digitises sound and transmits it to the implant. An electric stimulus from the implant mimics the change in electrical potential normally caused by the movement of stereocilia in the cochlea when a sound occurs. This change generates an impulse along the auditory nerve to the brain resulting in perception of sound.

CIs are available in the UK to people who have profound hearing loss. The improvement of CI technology means individuals with less significant losses, or profound losses at only some pitches may now benefit from a CI over a hearing aid. Patients having useful residual hearing has led to interest in better preserving that hearing during surgery. Thus allowing benefit from traditional acoustic amplification in addition to electrical stimulation from the implant.

The investigators propose recording a measurement via the implant during surgery and at audiology appointments called a cochlear microphonic using a technique called electrocochleography (ECochG). This is essentially recording the electrical signal generated by the movement of hair cells in the cochlea in response to a sound. It is hypothesised that reduction of this signal during implantation may correspond to cochlea damage occurring and that with development this signal might be useful feedback for surgeons. The signal is known to be correlated to actual hearing ability so a better understanding of this may allow us to fit the acoustic amplification portion of implants in individuals who are unable to respond reliably to a normal hearing test.

The purpose of this study is a pilot to assess the correlation between observed changes in this signal during surgery and residual hearing loss post-operatively and the degree correlation between recordings of this signal post-operatively and actual hearing test results.

ELIGIBILITY:
Inclusion Criteria:

* Meets normal candidacy requirements for cochlear implantation
* At least 1 year of age at time of consent being given
* Patent cochlea as verified by CT or MRI scan
* No cochlear abnormality that might prevent insertion of the electrode array
* Measurable residual hearing in the ear to be implanted
* No additional complex needs that would prevent study procedures or normal clinical follow-up protocol being followed
* AB Implant selected by patient or MDT
* Written informed consent obtained

Exclusion Criteria:

* Medically complex cases where minimal duration of surgery is required

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-01-24 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Cochlear Microphonic Amplitude (micro volts) via Electrocochleography during Cochlear Implant Insertion | 1 Year
  Cochlear Microphonic amplitude from real time electrocochleography using the apical cochlear implant electrode during implant insertion.
Cochlear Microphonic Amplitude (micro volts) via Electrocochleography during post-operative audiological appointments | 1 Year
  Cochlear Microphonic amplitude recorded from varying electrodes and at varying frequencies post-insertion during each follow-up appointment for the first year.

SECONDARY OUTCOMES:
ECochG Correlations | 1 Year
  Correlations between Intra and Post-operative cochlear microphonic amplitudes and other normal clinical measures (Impedance, eCAP, PTA, Speech)

CONTACTS AND LOCATIONS:
Overall Officials: Terry B Nunn, MSc, Principal Investigator — Head of Audiology and Consultant Clinical Scientist; Dan Jiang, PhD FRCS, Study Chair — Professor of Otology and Auditory Implantation Surgery.
Locations (1):
- Hearing Implant Centre, Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dalbert A, Pfiffner F, Hoesli M, Koka K, Veraguth D, Roosli C, Huber A. Assessment of Cochlear Function during Cochlear Implantation by Extra- and Intracochlear Electrocochleography. Front Neurosci. 2018 Jan 26;12:18. doi: 10.3389/fnins.2018.00018. eCollection 2018. PMID 29434534
- [Background] Pienkowski M, Adunka OF, Lichtenhan JT. Editorial: New Advances in Electrocochleography for Clinical and Basic Investigation. Front Neurosci. 2018 May 8;12:310. doi: 10.3389/fnins.2018.00310. eCollection 2018. No abstract available. PMID 29867322
- [Background] Koka K, Saoji AA, Litvak LM. Electrocochleography in Cochlear Implant Recipients With Residual Hearing: Comparison With Audiometric Thresholds. Ear Hear. 2017 May/Jun;38(3):e161-e167. doi: 10.1097/AUD.0000000000000385. PMID 27879487
- [Background] O'Connell BP, Holder JT, Dwyer RT, Gifford RH, Noble JH, Bennett ML, Rivas A, Wanna GB, Haynes DS, Labadie RF. Intra- and Postoperative Electrocochleography May Be Predictive of Final Electrode Position and Postoperative Hearing Preservation. Front Neurosci. 2017 May 29;11:291. doi: 10.3389/fnins.2017.00291. eCollection 2017. PMID 28611574
- [Background] Mandala M, Colletti L, Tonoli G, Colletti V. Electrocochleography during cochlear implantation for hearing preservation. Otolaryngol Head Neck Surg. 2012 May;146(5):774-81. doi: 10.1177/0194599811435895. Epub 2012 Jan 30. PMID 22291043
- [Derived] Soulby A, Connor S, Jiang D, Nunn T, Boyle P, Pai I. Establishing Reproducibility and Correlation of Cochlear Microphonic Amplitude to Implant Electrode Position Using Intraoperative Electrocochleography and Postoperative Cone Beam Computed Tomography. Ear Hear. 2021 Sep/Oct;42(5):1263-1275. doi: 10.1097/AUD.0000000000001010. PMID 33813521